CLINICAL TRIAL: NCT05233683
Title: Caudal Block Versus Dorsal Penile Nerve Block Plus Ring Block for Pain Management of Different Surgical Techniques of Circumcision in Infants and Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Mansoor Aqil, Professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-21-5965
Record Dates: First submitted 2021-10-22; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia; Anesthesia, Local; Analgesia; Pediatric ALL; Pain, Postoperative; Pain, Acute
MeSH Terms: conditions — Agnosia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pain, Postoperative; Acute Pain | interventions — Circumcision, Male

STUDY DESIGN:
Intervention Model Description: All patients will receive general anesthesia. Patients will be randomly allocated to one of 4 arms of the study:
  * Group 1 will receive are caudal block (CB) and circumcision with Plastibell,
  * Group 2 will receive CB and circumcision with conventional dissection method (CDM),
  * Group 3 will receive dorsal penile block (DPNB) and ring block (RB) and circumcision with Plastibell, and
  * Group 4 will receive DPNB+ RB and circumcision with CDM.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Caudal block and circumcision with Plastibell, (Experimental): Caudal block will be performed with 0.75ml/kg of 0.25% bupivacaine containing 1 mic/kg dexmedetomidine. Circumcision will be done using plastibell. Paracetamol suppository will also be inserted per rectum in the dose of 15 mg/kg before the start of surgery. The surgery will be started 10 minutes after block placement to allow adequate time for the block to be effective.
  Interventions: Drug: Caudal block; Procedure: Circumcision with Plastibell
- Caudal block and circumcision with conventional dissection method (Experimental): Caudal block will be performed with 0.75ml/kg of 0.25% bupivacaine containing 1 mic/kg dexmedetomidine. Circumcision will be done using the conventional dissection method. Paracetamol suppository will also be inserted per rectum in the dose of 15 mg/kg before the start of surgery. The surgery will be started 10 minutes after block placement to allow adequate time for the block to be effective.
  Interventions: Drug: Caudal block; Procedure: Conventional Dissection Method
- Dorsal penile nerve block plus ring block and circumcision with Plastibell (Active Comparator): Dorsal penile nerve block plus ring block with 0.25% bupivacaine. Circumcision will be done using plastibell.
  Interventions: Drug: Dorsal penile nerve block plus ring block; Procedure: Circumcision with Plastibell
- Dorsal penile nerve block plus ring block and circumcision with conventional dissection method (Active Comparator): Dorsal penile nerve block plus ring block with 0.25% bupivacaine. Circumcision will be done using the conventional dissection method
  Interventions: Drug: Dorsal penile nerve block plus ring block; Procedure: Conventional Dissection Method

INTERVENTIONS:
Drug: Caudal block — Caudal block will be performed in lateral position with 0.25% bupivacaine in the dose of 0.75 ml/kg containing 1 mic/kg dexmedetomidine. The patients will be turned back to the supine position after the block placement and the head of the patient will be placed in the neutral position. Paracetamol suppository will also be inserted per rectum in the dose of 15 mg/kg before the start of surgery. The surgery will be started 10 minutes after block placement to allow adequate time for the block to be effective.
  Arms: Caudal block and circumcision with Plastibell,; Caudal block and circumcision with conventional dissection method
Drug: Dorsal penile nerve block plus ring block — It will be performed with the child in the supine position. Following skin preparation and palpation of the arch of the lower border of the symphysis pubis, the base of the penis will be gently pulled down, and a 25-G needle will be inserted at 10 and 2.0 "O" clock position to a depth of 0.25-0.5 cm (under Bucks' fascia) and 1 ml + 0.1ml X weight of the patient) of local anesthetic (0.25% bupivacaine) will be injected at each point after negative aspiration and then RB will be done in the form of a circumferential subcutaneous ring at the level of the base of the penis. Paracetamol suppository will also be inserted per rectum in the dose of 15 mg/kg before the start of surgery. The surgery will be started 10 minutes after block placement to allow adequate time for the block to be effective.
  Arms: Dorsal penile nerve block plus ring block and circumcision with Plastibell; Dorsal penile nerve block plus ring block and circumcision with conventional dissection method
Procedure: Circumcision with Plastibell — Circumcision with Plastibell
  Arms: Caudal block and circumcision with Plastibell,; Dorsal penile nerve block plus ring block and circumcision with Plastibell
Procedure: Conventional Dissection Method — Conventional Dissection Method
  Arms: Caudal block and circumcision with conventional dissection method; Dorsal penile nerve block plus ring block and circumcision with conventional dissection method

SUMMARY:
Circumcision is one of the most commonly performed operations in the pediatric population and is a painful procedure. Circumcision is performed with two popular techniques, Plastibell and conventional dissection method (CDM). For intra-operative (OP) and post-OP pain relief, two commonly used local anesthetic techniques are caudal block (CB) and dorsal penile block (DPNB) plus ring block (RB) at the base of the penis. There are very few randomized controlled trials comparing these two methods of intra-OP and post-OP pain relief, for different surgical techniques and there is a lack of well-conducted studies comparing the quality of analgesia, need for rescue analgesia in the early post-OP period, complications, and parental satisfaction comparing these blocks. Furthermore, there is a lot of contradiction in the literature regarding the duration of analgesia produced with these techniques.

DETAILED DESCRIPTION:
Circumcision is one of the most commonly performed operations in the paediatric population and is a painful procedure. Circumcision is performed with two popular techniques, Plastibell and conventional dissection method. Two anesthetic techniques are commonly used for intra-operative (OP) and post-OP pain relief i.e CB and DPNB+RB at the base of the penis. Addition of dexmedetomidine to bupivacaine prolongs duration of analgesia of CB. Both anaesthesia techniques of pain relief have certain advantages and disadvantages and the superiority of any technique over the other has not been established.

There are very few randomized controlled trials comparing these two methods of intra-OP and post-OP pain relief, for different surgical techniques of circumcision and there is a lack of well-conducted studies comparing the quality of analgesia, need for rescue analgesia in the early post-OP period, complications, and parental satisfaction comparing these blocks. Furthermore, there is a lot of contradiction in the literature regarding the duration of analgesia produced with these techniques.

Poorly treated postoperative pain leads to fatigue and metabolic, endocrine, and immunological changes can lead to prolonged convalescence following surgery and is traumatic to the pediatric patients and their parents. In this study, the investigators planned to compare the two most popular methods of pain relief during and after circumcision, along with parents' satisfaction.

This research will guide the anesthetists regarding the selection of appropriate techniques of intra-OP and post-OP analgesia and in light of intra and post-OP data; and parents' satisfaction.

In this prospective randomized study the investigators plan to compare the quality of intra and post OP analgesia and the duration of post-OP analgesia produced by CB and DPNB +RB, need of rescue analgesia with both of the techniques of surgery, intra-OP hemodynamic variations, residual motor block, and adverse effects and parents' satisfaction with both of the anesthesia and the surgical techniques.

Research Objectives:

To evaluate and compare the intra and post-OP pain relief under CB and DPNB plus RB in pediatric patients undergoing circumcision with different surgical techniques and assessment of parents' satisfaction

This study may guide the anesthetists for the selection of appropriate techniques of intra and post-OP analgesia and their complications for different surgical techniques of circumcision and also about parent's satisfaction with the anesthetic technique.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy,
2. Male,
3. Ages 3 months to 4 years,
4. Scheduled for circumcision for various indications under GA.

Exclusion Criteria:

1. Patients with bleeding or clotting disorders
2. Patients with hypospadias, other penile or sacral anomalies
3. Patients weight <3kg.
4. Allergy to Local Anesthetic
5. Infection at the site of block
6. Pre-existing spinal or neurological disease
7. Pain medication within the previous 48 hours

Ages: 3 Months to 4 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Patient eligibility is based on gender identity
Enrollment: 120 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of analgesia using FLACC Scale | First 12 hours after surgery/intervention (circumcision)
  Postoperatively in the PACU, the child will be observed in the recovery room by a senior nurse blinded to the anesthetic technique and the FLACC score will be used for pain assessment (copy attached). The FLACC scale is a uni-dimensional behavioral pain assessment instrument to measure pain in young children in the post-OP period. It includes five items (Face, Leg, Activity, Cry, and Consolability) and has good inter-rater reliability (Kappa 0.52-0.82), as well as good content and convergent validity. The scale is scored in a range of 0-10 with 0 = no pain and 10 = severe pain. The FLACC is reliable in critically ill young children. The severity of pain will be classified using the total score 0=no pain, and 10= severe pain. I.V fentanyl will be administered in the dose of 0.5 mic/kg if the pain score is >5 and the dose will be repeated if the FLACC score persisted >5 after five minutes.
Duration of analgesia | First 12 hours after surgery/intervention (circumcision)
  To compare the duration of post-OP analgesia produced by CB and DPNB plus RB in children undergoing circumcision with two different surgical techniques.

SECONDARY OUTCOMES:
Number of participants that needed rescue analgesia | first 12 hours after surgery (circumcision)
  Number of participants that needed rescue analgesia in PACU and ward
Motor block score | first 12 hours after surgery (circumcision)
  Motor block score will be recorded (0=spontaneous movements of hips, knees and ankles, 1=movements of knees and ankles but no movements of hips, 2=only movements of ankles, and 3=no movements of lower limbs).
Blood pressure (mm/Hg) | during the surgery (from start time to end time of circumcision)
  Patients will receive fentanyl 0.5 mic/kg, if at any stage HR or BP increased 25% more than baseline value and the total dose of rescue analgesia received intra-operatively will be recorded.
Heart rate (beats/min) | during the surgery (from start time to end time of circumcision)
  Patients will receive fentanyl 0.5 mic/kg, if at any stage HR or BP increased 25% more than baseline value and the total dose of rescue analgesia received intra-operatively will be recorded.
Time to discharge from PACU | First 12 hours after surgery (circumcision)
  Amount of time the patient stays in PACU after the surgery. This will be a continuous variable (time).
Number of patients with infection | First 5 days after surgery (circumcision)
  Number of patients experiencing infection at site of circumcision. It will be recorded as yes/no.
Number of patients experiencing urinary retention | First 12 hours after surgery (circumcision)
  Measured as: no urine output after intervention.
Number of Participants with sedation | First 12 hours after surgery: assessed at 5, 15, and 30 minutes in PACU and hourly in the ward
  Sedation will be measured using the The Pasero Opioid-Induced Sedation Scale (POSS). POSS is a standardized approach to assessing opioid-induced sedation and instituting interventions. The POSS scores are S ("sleep, easy to arouse"), 1 ("awake and alert"), 2 ("slightly drowsy, easily aroused"), 3 ("frequently drowsy, arousable, drifts off to sleep during conversation"), and 4 ("somnolent, minimal, or no response to verbal or physical stimulation"). Scores of S, 1, or 2 are considered acceptable; the opioid dose may be increased if needed.
Number of Participants with nausea | First 12 hours after surgery: assessed at 5, 15, and 30 minutes in PACU and hourly in the ward
  Will be recorded as yes/no
Number of Participants with vomiting | First 12 hours after surgery: assessed at 5, 15, and 30 minutes in PACU and hourly in the ward
  Will be recorded as yes/no
Number of Participants with agitation | First 12 hours after surgery: assessed at 5, 15, and 30 minutes in PACU and hourly in the ward
  Will be recorded as yes/no
Number of Participants with penile hematoma | First 12 hours after surgery/intervention: assessed at 5, 15, and 30 minutes in PACU and hourly in the ward
  Will be recorded as yes/no
Total paracetamol doses administered | first 5 days after surgery (circumcision)
  Amount of paracetamol required by the patient for pain control

OTHER OUTCOMES:
Parents' satisfaction with pain relief using Likert Scale | First 5 days after surgery (circumcision)
  Parents' satisfaction with pain relief will be measured using a Likert Scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor Aqil, FCPS, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Rossi S, Buonocore G, Bellieni CV. Management of pain in newborn circumcision: a systematic review. Eur J Pediatr. 2021 Jan;180(1):13-20. doi: 10.1007/s00431-020-03758-6. Epub 2020 Aug 3. PMID 32748017
- [Background] Bawazir OA. A controlled trial of Gomco versus Plastibell for neonatal circumcisions in Saudi Arabia. Int J Pediatr Adolesc Med. 2020 Sep;7(3):132-135. doi: 10.1016/j.ijpam.2019.03.002. Epub 2019 Mar 21. PMID 33094142
- [Background] Jiang ZL, Sun CW, Sun J, Shi GF, Li H. Subcutaneous tissue-sparing dorsal slit with new marking technique: A novel circumcision method. Medicine (Baltimore). 2019 Apr;98(16):e15322. doi: 10.1097/MD.0000000000015322. PMID 31008987
- [Background] Weksler N, Atias I, Klein M, Rosenztsveig V, Ovadia L, Gurman GM. Is penile block better than caudal epidural block for postcircumcision analgesia? J Anesth. 2005;19(1):36-9. doi: 10.1007/s00540-004-0287-8. PMID 15674514
- [Background] Soltany S, Ardestanizadeh A. The study of the factors affecting the time of ring fall off in circumcision using Plastibell. J Family Med Prim Care. 2020 Jun 30;9(6):2736-2740. doi: 10.4103/jfmpc.jfmpc_1261_19. eCollection 2020 Jun. PMID 32984117
- [Background] O'Sullivan MJ, Mislovic B, Alexander E. Dorsal penile nerve block for male pediatric circumcision--randomized comparison of ultrasound-guided vs anatomical landmark technique. Paediatr Anaesth. 2011 Dec;21(12):1214-8. doi: 10.1111/j.1460-9592.2011.03722.x. PMID 22023417
- [Background] Wang X, Dong C, Beekoo D, Qian X, Li J, Shang-Guan WN, Jiang X. Dorsal Penile Nerve Block via Perineal Approach, an Alternative to a Caudal Block for Pediatric Circumcision: A Randomized Controlled Trial. Biomed Res Int. 2019 Mar 27;2019:6875756. doi: 10.1155/2019/6875756. eCollection 2019. PMID 31032356
- [Background] Teunkens A, Van de Velde M, Vermeulen K, Van Loon P, Bogaert G, Fieuws S, Rex S. Dorsal penile nerve block for circumcision in pediatric patients: A prospective, observer-blinded, randomized controlled clinical trial for the comparison of ultrasound-guided vs landmark technique. Paediatr Anaesth. 2018 Aug;28(8):703-709. doi: 10.1111/pan.13429. Epub 2018 Jul 23. PMID 30035357
- [Background] Heller GZ, Manuguerra M, Chow R. How to analyze the Visual Analogue Scale: Myths, truths and clinical relevance. Scand J Pain. 2016 Oct;13:67-75. doi: 10.1016/j.sjpain.2016.06.012. Epub 2016 Jul 27. PMID 28850536
- [Background] Chan KH, Shah A, Moser EA, Szymanski K, Whittam BM, Misseri R, Kaefer M, Rink R, Cain MP. Comparison of Intraoperative and Early Postoperative Outcomes of Caudal vs Dorsal Penile Nerve Blocks for Outpatient Penile Surgeries. Urology. 2018 Aug;118:164-171. doi: 10.1016/j.urology.2017.08.062. Epub 2017 Nov 6. PMID 29122625
- [Background] Panda A, Bajwa SJ, Sen S, Parmar SS. Penile block for paediatric urological surgery: A comparative evaluation with general anaesthesia. Indian J Urol. 2011 Oct;27(4):457-64. doi: 10.4103/0970-1591.91432. PMID 22279309
- [Background] Sandeman DJ, Reiner D, Dilley AV, Bennett MH, Kelly KJ. A retrospective audit of three different regional anaesthetic techniques for circumcision in children. Anaesth Intensive Care. 2010 May;38(3):519-24. doi: 10.1177/0310057X1003800317. PMID 20514962
- [Background] Yao Y, Yu C, Zhang X, Guo Y, Zheng X. Caudal and intravenous dexmedetomidine similarly prolong the duration of caudal analgesia in children: A randomized controlled trial. Paediatr Anaesth. 2018 Oct;28(10):888-896. doi: 10.1111/pan.13469. PMID 30302881
- [Background] Sharara-Chami R, Lakissian Z, Charafeddine L, Milad N, El-Hout Y. Combination Analgesia for Neonatal Circumcision: A Randomized Controlled Trial. Pediatrics. 2017 Dec;140(6):e20171935. doi: 10.1542/peds.2017-1935. Epub 2017 Nov 17. PMID 29150457
- [Background] Munevveroglu C, Gunduz M. Postoperative pain management for circumcision; Comparison of frequently used methods. Pak J Med Sci. 2020 Jan-Feb;36(2):91-95. doi: 10.12669/pjms.36.2.505. PMID 32063938
- [Background] Cyna AM, Middleton P. Caudal epidural block versus other methods of postoperative pain relief for circumcision in boys. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD003005. doi: 10.1002/14651858.CD003005.pub2. PMID 18843636
- [Background] Sinkey RG, Eschenbacher MA, Walsh PM, Doerger RG, Lambers DS, Sibai BM, Habli MA. The GoMo study: a randomized clinical trial assessing neonatal pain with Gomco vs Mogen clamp circumcision. Am J Obstet Gynecol. 2015 May;212(5):664.e1-8. doi: 10.1016/j.ajog.2015.03.029. Epub 2015 Mar 17. PMID 25794628
- [Background] Mehmood T, Azam H, Tariq M, Iqbal Z, Mehmood H, Shah SA. Plastibell Device Circumcision versus Bone Cutter Technique in terms of Operative Outcomes and Parent's Satisfaction. Pak J Med Sci. 2016 Mar-Apr;32(2):347-50. doi: 10.12669/pjms.322.9510. PMID 27182237
- [Background] Margetts L, Carr A, McFadyen G, Lambert A. A comparison of caudal bupivacaine and ketamine with penile block for paediatric circumcision. Eur J Anaesthesiol. 2008 Dec;25(12):1009-13. doi: 10.1017/S0265021508004833. Epub 2008 Jul 24. PMID 18652709
- [Background] Atasever AG, Ermis O, Demir BS, Kasali K, Karadeniz MS. Comparison of bupivacaine alone and in a combination with lidocaine for caudal block in patients undergoing circumcision: A historical cohort study. Turk J Urol. 2019 Nov 29;46(3):243-248. doi: 10.5152/tud.2019.19191. Print 2020 May. PMID 32401707
- [Background] Sottas CE, Anderson BJ. Dexmedetomidine: the new all-in-one drug in paediatric anaesthesia? Curr Opin Anaesthesiol. 2017 Aug;30(4):441-451. doi: 10.1097/ACO.0000000000000488. PMID 28537937
- [Background] Li S, Liu T, Xia J, Jia J, Li W. Effect of dexmedetomidine on prevention of postoperative nausea and vomiting in pediatric strabismus surgery: a randomized controlled study. BMC Ophthalmol. 2020 Mar 5;20(1):86. doi: 10.1186/s12886-020-01359-3. PMID 32138784
- [Background] Mahmoud M, Mason KP. Dexmedetomidine: review, update, and future considerations of paediatric perioperative and periprocedural applications and limitations. Br J Anaesth. 2015 Aug;115(2):171-82. doi: 10.1093/bja/aev226. PMID 26170346
- [Background] Bellon M, Le Bot A, Michelet D, Hilly J, Maesani M, Brasher C, Dahmani S. Efficacy of Intraoperative Dexmedetomidine Compared with Placebo for Postoperative Pain Management: A Meta-Analysis of Published Studies. Pain Ther. 2016 Jun;5(1):63-80. doi: 10.1007/s40122-016-0045-2. Epub 2016 Feb 10. PMID 26861737
- [Background] Mittino I, Sangalli M, Fabbri F, Sozzi F, Ghezzi M, Zanni G, Cestari A. Ischemia of the glans 24 hours after circumcision: A case report and therapeutic solution. Urologia. 2018 Nov;85(4):174-176. doi: 10.1177/0391560318761288. Epub 2018 Mar 26. PMID 30426879
- [Background] Ozen V, Yigit D. A comparison of the postoperative analgesic effectiveness of low dose caudal epidural block and US-guided dorsal penile nerve block with in-plane technique in circumcision. J Pediatr Urol. 2020 Feb;16(1):99-106. doi: 10.1016/j.jpurol.2019.10.020. Epub 2019 Oct 30. PMID 31759904